CLINICAL TRIAL: NCT04158141
Title: Phase III Randomized Trial of Pleurectomy/Decortication Plus Systemic Therapy With or Without Adjuvant Hemithoracic Intensity-Modulated Pleural Radiation Therapy (IMPRINT) for Malignant Pleural Mesothelioma (MPM)
Brief Title: Testing the Addition of Targeted Radiation Therapy to Surgery and the Usual Chemotherapy Treatment (Pemetrexed and Cisplatin [or Carboplatin]) for Stage I-IIIA Malignant Pleural Mesothelioma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Permanent Administrative Closure
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-LU006; NCI-2019-07141 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-LU006 (Other: NRG Oncology); NRG-LU006 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-12

CONDITIONS: Pleural Biphasic Mesothelioma; Pleural Epithelioid Mesothelioma; Stage I Pleural Malignant Mesothelioma AJCC v8; Stage IA Pleural Malignant Mesothelioma AJCC v8; Stage IB Pleural Malignant Mesothelioma AJCC v8; Stage II Pleural Malignant Mesothelioma AJCC v8; Stage IIIA Pleural Malignant Mesothelioma AJCC v8
Keywords: Mesothelioma; IMPRINT
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cerebral Decortication; Radiotherapy, Intensity-Modulated; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Step 1: chemotherapy, P/D: Step 2: no treatment) (Active Comparator): STEP 1: Patients who received allowed neoadjuvant systemic therapy before study entry undergo pleurectomy/decortication (P/D) within 4 to 8 weeks of systemic therapy. Otherwise, patients undergo P/D within 4 weeks of study entry followed within 4 to 8 weeks by four 21-day cycles of pemetrexed and cisplatin or carboplatin on day 1.
  STEP 2: Patients receive no treatment.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Decortication; Drug: Pemetrexed; Drug: Pemetrexed Disodium; Procedure: Pleurectomy
- Arm II (Step 1: chemotherapy, P/D, Step 2: IMRT/PBS) (Experimental): STEP 1: Same as Arm 1.
  STEP 2: Within 4-8 weeks from the end of Step 1 treatment, patients undergo 25-28 fractions of intensity modulated radiation therapy (IMRT) or pencil beam scanning (PBS) proton therapy 5 days/week over 6 weeks.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Decortication; Radiation: Intensity-Modulated Radiation Therapy; Drug: Pemetrexed; Drug: Pemetrexed Disodium; Radiation: Pencil beam scanning proton therapy; Procedure: Pleurectomy

INTERVENTIONS:
Drug: Carboplatin — Intravenously
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Intravenously
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Decortication — Undergo decortication
Radiation: Intensity-Modulated Radiation Therapy — Daily fractions
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: Arm II (Step 1: chemotherapy, P/D, Step 2: IMRT/PBS)
Drug: Pemetrexed — Intravenously
  Other Names: MTA; Multitargeted Antifolate
Drug: Pemetrexed Disodium — Intravenously
  Other Names: Alimta; Almita; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Radiation: Pencil beam scanning proton therapy — Daily fractions
  Other Names: PBS proton therapy; intensity modulated proton therapy
  Arms: Arm II (Step 1: chemotherapy, P/D, Step 2: IMRT/PBS)
Procedure: Pleurectomy — Undergo pleurectomy
  Other Names: Excision of Pleura

SUMMARY:
This trial studies how well the addition of targeted radiation therapy to surgery and the usual chemotherapy treatment works for the treatment of stage I-IIIA malignant pleural mesothelioma. Targeted radiation therapy such as intensity-modulated radiation therapy or pencil beam scanning uses high energy rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as pemetrexed, cisplatin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving targeted radiation therapy in addition to surgery and chemotherapy may work better than surgery and chemotherapy alone for the treatment of malignant pleural mesothelioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To detect an improvement in overall survival with the addition of adjuvant hemithoracic intensity-modulated pleural radiation therapy (IMPRINT) to surgery and chemotherapy compared to surgery and chemotherapy alone.

SECONDARY OBJECTIVES:

I. To determine local failure-free survival, distant-metastases-free survival, and progression-free survival with the addition of adjuvant hemithoracic IMPRINT to surgery and chemotherapy compared to surgery and chemotherapy alone.

II. To evaluate the treatment-related toxicities in both arms per Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

III. To detect a clinically meaningful 10-point change in global health status mean scores at 9 months after randomization with the addition of adjuvant IMPRINT as compared to surgery and chemotherapy alone.

EXPLORATORY OBJECTIVES:

I. To evaluate the degree of under-staging, concordant and upstaging between centrally reviewed clinical staging (based on positron emission tomography (PET), computed tomography (CT) and/or magnetic resonance imaging (MRI)) and pathologic staging.

II. To identify immunologic and pathologic biomarkers as predictors of response and potential targets for future combination trials.

III. To determine the magnitude of radiation dose escalation to gross residual disease based on combined modality imaging and associated local control rates with dose-painting intensity-modulated radiation therapy (IMRT).

IV. To determine the rate of R0/R1 and R2 resections, and type of procedures (extended pleurectomy/decortication [P/D], P/D and partial pleurectomy).

V. To evaluate the trajectory of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-Q30) and lung cancer specific module (LC13) symptoms in patients treated with IMPRINT by comparing the proportion of patients who respond with "quite a bit" or "very much" LC13 symptoms at 9-12 months post-randomization compared to at 3 months post-randomization.

VI. To evaluate changes in health-related quality of life, functional domains, and symptoms over time with the addition of adjuvant IMPRINT as compared to surgery and chemotherapy alone.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

PRIOR TO STEP 1 REGISTRATION - ALL PATIENTS

* Pathologically (histologically or cytologically) confirmed diagnosis of epithelioid or biphasic malignant pleural mesothelioma (MPM)
* Imaging proof of clinical stage (American Joint Committee on Cancer [AJCC] 8th edition) I-IIIA MPM by PET/CT;

  * Diagnostic volumetric CT scan of the chest is preferred; however, the CT portion of the PET/CT may be used if CT imaging is of diagnostic quality
* MPM is amenable to resection by P/D as determined by a thoracic surgeon
* History/physical examination within 42 days prior to Step 1 Registration
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 within 42 days prior to Step 1 Registration
* Required Initial Laboratory Values prior to study entry (must be at least 14 days after last infusion of pre-study entry neoadjuvant therapy, if given):

  * Absolute neutrophil count ≥1500 cells/mm3;
  * Platelets ≥100,000 cells/mm3;
  * Hemoglobin ≥ 8.0 g/dL;
  * Serum total bilirubin ≤ 1.5 X ULN (upper limit of normal);
  * Aspartate transferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine transaminase (ALT) (serum glutamic-oxaloacetic transaminase (SGPT)) ≤ 3.0 X ULN;
  * Creatinine clearance ≥45 mL/min by the Cockcroft-Gault (C-G) equation
* Negative serum pregnancy test within 14 days of Step 1 Registration for women of childbearing potential
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Note: HIV testing is not required for eligibility for this protocol.
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

PRIOR TO STEP 1 REGISRATION - PATIENTS WHO RECEIVED SYSTEMIC THERAPY BEFORE STUDY ENTRY

* The following systemic therapy and immunotherapy combinations are permissible: 1) cisplatin/carboplatin + pemetrexed; 2) cisplatin/carboplatin + pemetrexed + anti-PD-1/L1 agents; and 3) ipilimumab/nivolumab.
* Patients must have received at least 2 cycles of neoadjuvant systemic therapy

PRIOR TO STEP 2 RANDOMIZATION - ALL PATIENTS

* No evidence of progression as defined by PET/CT within 30 days prior to Step 2 randomization.
* Patients must have received at least 2 cycles of systemic therapy and undergone a pleurectomy/decortication with the goal of macroscopic complete resection;
* ECOG Performance Status 0-1 within 30 days prior to Step 2 Randomization
* History/physical examination within 30 days prior to Step 2 Randomization

Exclusion Criteria:

PRIOR TO STEP 1 REGISTRATION - ALL PATIENTS

* Pregnancy or women who are breastfeeding and unwilling to discontinue.
* Participants of childbearing potential (participants who may become pregnant or who may impregnate a partner) unwilling to use highly effective contraceptives during and for six months after end of treatment because the treatment in this study may be significantly teratogenic.
* Diagnosis of sarcomatoid mesothelioma
* Severe, active co-morbidity defined as follows:

  * New York Heart Association (NYHA) class III or IV heart failure
  * Chronic obstructive pulmonary disease (COPD) requiring chronic oral steroid therapy of > 10 mg prednisone daily or equivalent at the time of registration. Inhaled corticosteroids are allowed;
  * Unstable angina requiring hospitalization and/or transmural myocardial infarction within the last 3 months;
  * Interstitial lung disease;
  * Hemodialysis or peritoneal dialysis;
  * Concurrent active malignancy (with the exception of current or prior non-melanomatous skin cancer or low-grade malignancies followed observantly for which treatment has not or does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen)

    * If evidence of disease < 3 years, institution must consult with the principal investigator, Andreas Rimner, Doctor of Medicine (MD)
  * Hepatic impairment defined by ChildPugh class (ChildPugh class B & C);

    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy within 30 days prior to registration, if indicated. Note: HBV viral testing is not required for eligibility for this protocol
    * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load within 30 days prior to registration
  * • Active lung infection requiring IV antibiotics
  * Patients on immunosuppressive therapy, for example history of organ or bone marrow transplant or other hematologic disorders that are expected to compromise life expectancy or tolerance of treatment;
* Prior nephrectomy on the contralateral side of MPM
* Ipsilateral thoracic electronic implant, e.g. pacemaker, defibrillator, unless switched to the contralateral side prior to initiation of radiation therapy (RT)
* Prior thoracic radiation therapy (patients with prior thoracic RT cannot be planned to 50-60 Gy without exceeding normal tissue constraints)
* Use of bevacizumab or other antiangiogenic therapy to treat current mesothelioma (due to potential for increased complications from local therapy).
* For patients who received neoadjuvant systemic therapy prior to study entry, surgery planned to occur greater than 8 weeks following neoadjuvant systemic therapy

PRIOR TO STEP 2 RANDOMIZATION - ALL PATIENTS

* Supplemental oxygen use
* Third space fluid that cannot be controlled by drainage or insufficient lung expansion after P/D (this prevents targeting the pleura without exceeding normal tissue constraints)
* Prior intrapleural therapy (i.e. intrapleural chemotherapy, photodynamic therapy); pleurodesis is permitted
* Bulky residual disease in the major fissure preventing pleural IMRT
* Patients who have undergone extrapleural pneumonectomy
* Patients with active infection that requires systemic I.V. antibiotics, antiviral, or antifungal treatments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Rimner, MD, Principal Investigator — NRG Oncology
Locations (27):
- United States (26):
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson in The Woodlands, Conroe, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Swedish Medical Center-First Hill, Seattle, Washington
- The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Registered, Not Yet Randomized: All patients are on Step 1 before being randomized to Step 2.
  STEP 1: Patients who received allowed neoadjuvant systemic therapy before study entry undergo pleurectomy/decortication (P/D) within 4 to 8 weeks of systemic therapy. Otherwise, patients undergo P/D within 4 weeks of study entry followed within 4 to 8 weeks by four 21-day cycles of pemetrexed and cisplatin or carboplatin on day 1.
Period: Step 1: Registration
Arm/Group | Registered, Not Yet Randomized | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Started | 16 | 0 | 0
Eligible (Step 1) | 16 | 0 | 0
Completed (Patients continuing to Step 2. Patients must have received at least 2 cycles of systemic therapy and undergone a pleurectomy/decortication with the goal of macroscopic complete resection; Within 30 days prior to Step 2 randomization: no evidence of progression, ECOG Performance Status 0-1, history/physical examination occurs.) | 11 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Does not meet requirements for Step 2 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Study terminated immediately after patient enrolled | 2 | 0 | 0
Period: Step 2: Randomization
Arm/Group | Registered, Not Yet Randomized | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Started | 0 | 5 | 6
Eligible (Step 2) | 0 | 5 | 6
Completed (Randomized patients contributing data to results are considered to have completed Step 2.) | 0 | 5 | 6
Not Completed | 0 | 0 | 0
Period: Step 2: As-treated Population
Arm/Group | Registered, Not Yet Randomized | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Started (These are the randomized patients grouped to treatment arm by the treatment they *received* rather than the treatment they were assigned. This population is used only for the single adverse event outcome measure.) | 0 | 6 | 4
Completed | 0 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Not randomized: Eligible registered patients who did not continue to Step 2 (randomization).
  Arm 1 and Arm 2: Eligible randomized patients.
Groups:
- Step 1 Only: Patients that did not continue to Step 2 (were not randomized). STEP 1: Patients who received allowed neoadjuvant systemic therapy before study entry undergo pleurectomy/decortication (P/D) within 4 to 8 weeks of systemic therapy. Otherwise, patients undergo P/D within 4 weeks of study entry followed within 4 to 8 weeks by four 21-day cycles of pemetrexed and cisplatin or carboplatin on day 1.
- Total: Total of all reporting groups
Arm/Group | Step 1 Only | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS) | Total
Number analyzed (Participants) | 5 | 5 | 6 | 16
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 0 | 1 | 1 | 2
  50 - 59 years | 0 | 2 | 1 | 3
  60 - 69 years | 1 | 1 | 2 | 4
  ≥ 70 years | 4 | 1 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 5 | 2 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status at Registration [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 3 | 2 | 2 | 7
    1 | 2 | 3 | 4 | 9
Cell type [Count of Participants; unit: Participants]
  Biphasic mesothelioma | 2 | 1 | 1 | 4
  Epithelioid | 3 | 4 | 5 | 12
Macroscopic complete resection in Step 1 [Count of Participants; unit: Participants] — Population: This is only a baseline characteristic for Step 2, because surgery occurs during Step 1.
  Participants
    number analyzed (Participants) | 0 | 5 | 6 | 11
    R0 (Complete resection) |  | 1 | 3 | 4
    R1 (Macroscopically complete resection) |  | 3 | 3 | 6
    R2 (Resection that leaves gross tumor behind) |  | 1 | 0 | 1
Yearly procedure volume at the patient's treatment center [Count of Participants; unit: Participants] — The yearly number of pleurectomy/decortication procedures performed at the treatment center where the patient underwent this procedure. This data is only a reported baseline measure for Step 2. Population: This data is only a reported baseline measure for Step 2.
  Participants
    < 10 pleurectomy/decortations: number analyzed (Participants) | 0 | 5 | 6 | 11
    < 10 pleurectomy/decortations |  | 1 | 2 | 3
    ≥ 10 pleurectomy/decortations: number analyzed (Participants) | 0 | 5 | 6 | 11
    ≥ 10 pleurectomy/decortations |  | 4 | 4 | 8
Pathologic AJCC Stage [Count of Participants; unit: Participants] — Overall cancer stage per American Joint Committee on Cancer (AJCC) 8th ed. combines tumor (T), regional lymph node (N), and distant metastasis (M) staging to determine an overall stage of 0, I, II, III, or IV, ranging from least to most advanced, respectively, with patients within the same stage sharing a similar prognosis. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. The higher the number after the N, the greater the involvement of regional lymph nodes. M0 indicates no distant metastasis.
  Participants
    IA (T1N0M0) | 0 | 3 | 0 | 3
    IIA (T2bN0M0) | 2 | 1 | 4 | 7
    IIB (T[1-2]N1M0,T3N0M0) | 2 | 1 | 1 | 4
    IIIA (T[1-2]N2M0) (T3N1M0) (T4N[0-1]M0) | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was to be estimated by the Kaplan-Meier method and arms were to be compared using a log-rank test. Analysis was to occur when at least 105 deaths had been reported. Given the small number of participants due to early study closure, only the number of patients last reported to be alive at time of study termination is reported.
Time Frame: Randomization to the date of death or last follow-up. Maximum follow-up time from randomization was 25 months.
Population: Randomized patients
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment): [Intent-to-treat]
  STEP 1 (all patients): Patients who received allowed neoadjuvant systemic therapy before study entry undergo pleurectomy/decortication (P/D) within 4 to 8 weeks of systemic therapy. Otherwise, patients undergo P/D within 4 weeks of study entry followed within 4 to 8 weeks by four 21-day cycles of pemetrexed and cisplatin or carboplatin on day 1.
  STEP 2 (randomized): Patients receive no treatment.
- Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS): [Intent-to-treat]
  STEP 1 (all patients): Same as Arm 1.
  STEP 2 (randomized): Within 4-8 weeks from the end of Step 1 treatment, patients undergo 25-28 fractions of intensity modulated radiation therapy (IMRT) or pencil beam scanning (PBS) proton therapy 5 days/week over 6 weeks.
Arm/Group | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Number analyzed (Participants) | 5 | 6
Participants | 5 | 4

2. Secondary Outcome: Local-failure-free Survival (LFFS)
Description: Local failure is defined as local enlargement (LE) or local failure (LF) tumor response, marginal failure (MF), or death. LFFS was to be estimated by the Kaplan-Meier method and arms compared by log-rank test. Analysis was to occur when at least 105 deaths had been reported. Given the small number of participants due to early study closure, only the number of patients last reported to be alive without failure at time of study termination is reported, and no statistical testing was done.
  LE: ≥ 20% increase in the largest diameter (LD) of target lesion from the smallest LD recorded since the treatment start; based on computed tomography (CT) scan.
  LF: Progression of pleural tumor thickness or appearance of a site of pleural thickness > 5 mm in the site of treated tumor.
  MF: The appearance of a new measurable site of pleural tumor > 5mm within the treated site or enlarging tumor dimensions corresponding to a 20% increase in LD compared to initial appearance on imaging evaluation.
Time Frame: From randomization to local failure, death, or last follow-up, whichever occurs first. Maximum follow-up was 25 months.
Population: Randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Number analyzed (Participants) | 5 | 6
Participants | 3 | 3

3. Secondary Outcome: Distant-metastases-free Survival (DMFS)
Description: Distant failure (DF) is defined as the appearance of cancer deposits characteristic of metastatic dissemination from mesothelioma. DMFS was to be estimated by the Kaplan-Meier method and arms were to be compared using a log-rank test. Analysis was to occur when at least 105 deaths had been reported. Given the small number of participants due to early study closure, only the number of patients last reported to be alive without failure at time of study termination is reported, and no statistical testing was done.
Time Frame: From randomization to distant failure, death, or last follow-up, whichever occurs first. Maximum follow-up was 25 months.
Population: Randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Number analyzed (Participants) | 5 | 6
Participants | 5 | 2

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined as LE, LF, MF, DF, or death. PFS was to be estimated by the Kaplan-Meier method and arms compared by log-rank test. Analysis was to occur when ≥ 105 deaths had been reported. Given the small number of participants due to early study closure, only the number of patients last reported to be alive without progression at study termination is reported, and no statistical testing was done.
  LE: ≥ 20% increase in the largest diameter (LD) of target lesion from the smallest LD recorded since the treatment start; based on CT scan.
  LF: Progression of pleural tumor thickness or appearance of a site of pleural thickness > 5 mm in the site of treated tumor.
  MF: The appearance of a new measurable site of pleural tumor > 5mm within the treated site or enlarging tumor dimensions corresponding to a 20% increase in LD compared to initial appearance on imaging evaluation.
  DF: The appearance of cancer deposits characteristic of metastatic dissemination
Time Frame: From randomization to first progression, death, or last follow-up, whichever occurs first. Maximum follow-up was 25 months.
Population: Randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Number analyzed (Participants) | 5 | 6
Participants | 3 | 2

5. Secondary Outcome: Number of Patients With Grade 3 or Higher Treatment-related Adverse Event After Randomization
Description: Common Terminology Criteria for Adverse Events (version 5.0) grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Adverse events reported as possibly, probably, or definitely related to treatment are considered to be treatment-related adverse events.
Time Frame: From randomization to death or last follow-up. Maximum follow-up time was 25 months.
Population: Randomized patients who received protocol treatment and were assessed for adverse events. Arms determined by Step 2 treatment received (as-treated).
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment): [As-treated]
  STEP 1 (all patients): Patients who received allowed neoadjuvant systemic therapy before study entry undergo pleurectomy/decortication (P/D) within 4 to 8 weeks of systemic therapy. Otherwise, patients undergo P/D within 4 weeks of study entry followed within 4 to 8 weeks by four 21-day cycles of pemetrexed and cisplatin or carboplatin on day 1.
  STEP 2 (randomized): Patients receive no treatment.
- Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS): [As-treated]
  STEP 1 (all patients): Same as Arm 1.
  STEP 2 (randomized): Within 4-8 weeks from the end of Step 1 treatment, patients undergo 25-28 fractions of intensity modulated radiation therapy (IMRT) or pencil beam scanning (PBS) proton therapy 5 days/week over 6 weeks.
Arm/Group | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Number analyzed (Participants) | 6 | 4
Participants | 0 | 1

6. Secondary Outcome: Change From Randomization to 9 Months in Global Heath Status (GHS) Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: Global Health Status is calculated from two questions on the EORTC QLQ-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best).
Time Frame: Randomization and 9 months
Population: No patients had both baseline and 9-month data, therefore change from baseline could not be calculated for any patient.
Arm/Group | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Proportion of Patients With Under-staging, Concordant and Upstaging Between Centrally-reviewed Clinical Staging and Pathologic Staging
Description: For each subject, the centrally-reviewed clinical staging (based on positron emission tomography, computed tomography and/or magnetic resonance imaging) will be compared with pathologic staging to determine whether it is under-staging (clinical staging is more extensive than pathologic staging), concordant (clinical staging is same as pathologic staging), or upstaging (clinical staging is less extensive than pathologic staging).
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Association Between Radiation Dose to Gross Residual Disease and Local Control
Description: Gross residual disease and local failure will be analyzed as competing risk data (death without gross residual disease or death without local failure as the respective competing event). Association between radiation dose to gross residual disease and local failure will be evaluated similarly in multivariable analyses using Fine-Gray regression model.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Rate of R0/R1 and R2 Resections, by Type of Procedures (Extended Pleurectomy/Decortication (P/D), P/D and Partial Pleurectomy)
Description: Proportions of R0/R1 and R2 resections, by type of procedures (extended pleurectomy/decortication (P/D), P/D and partial pleurectomy).
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Pre-randomization: From registration (Step 1) to randomization (Step 2). The timing of randomization could vary from approximately 8 weeks to 32 weeks, depending on several factors. Arm 1 and Arm 2: From randomization to last follow-up. Maximum follow-up was 25 months.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who started any protocol treatment and were assessed for adverse events.
Groups:
- Pre-randomization: All patients in Step 1.
  STEP 1 (all patients): Patients who received allowed neoadjuvant systemic therapy before study entry undergo pleurectomy/decortication (P/D) within 4 to 8 weeks of systemic therapy. Otherwise, patients undergo P/D within 4 weeks of study entry followed within 4 to 8 weeks by four 21-day cycles of pemetrexed and cisplatin or carboplatin on day 1.
Arm/Group | Pre-randomization | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/5 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 13/13 | 3/4 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-randomization (N=13) | Arm I (Step 1: Chemotherapy, P/D: Step 2: no Treatment) (N=4) | Arm II (Step 1: Chemotherapy, P/D, Step 2: IMRT/PBS) (N=6)
Anemia (Blood and lymphatic system disorders) | 5 | 0 | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0
Eye disorders - Other (Eye disorders) | 1 | 0 | 0
Watering eyes (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1
Chylous ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 8 | 0 | 2
Generalized edema (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Pain (General disorders) | 4 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 2 | 0 | 1
Investigations - Other (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysesthesia (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 16 subjects registered out of 140 planned (11 randomized out of 132 planned). Patients that were not randomized in Step 2 were not followed further. All data is reported as intent-to-treat except for the adverse event outcome measure, which is reported as as-treated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT04158141/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT04158141/ICF_001.pdf